CLINICAL TRIAL: NCT07321067
Title: Use of Immune Checkpoint Inhibitors in Patients With Advanced Hepatocellular Carcinoma : Efficacy and Outcomes
Acronym: ICIs
Status: Not yet recruiting | Type: Observational
Sponsor: Ahmed Karam Helmy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Karam Helmy, Use of immune checkpoint inhibitors in patients with advanced hepatocellular carcinoma : efficacy and outcomes, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med--25-12-8MD
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
Keywords: advanced hepatocellular carcinoma; immune checkpoint inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all patients diagnosed with advanced hepatocellular carcinoma eligible for ICIs

SUMMARY:
the Objectives of this study are:

• Primary Objective: To prospectively evaluate overall survival (OS), ICI-specific survival (OS-ICI), and progression-free survival (PFS) in patients with advanced HCC treated with immune checkpoint inhibitors.

the main question it aims to answer is: What are the clinical outcomes (overall survival, progression-free survival, and OS-ICIs) of immune checkpoint inhibitor therapy in patients with advanced hepatocellular carcinoma? Participants already taking immune checkpoint inhibitors as part of their regular medical care.

DETAILED DESCRIPTION:
Objectives • Primary Objective: To prospectively evaluate overall survival (OS), ICI-specific survival (OS-ICI), and progression-free survival (PFS) in patients with advanced HCC treated with immune checkpoint inhibitors.

• Secondary Objectives: To assess the incidence, type, and severity of irAEs. To identify clinical predictors of survival outcomes, including ALBI grade, prior LRT, SBRT or resection.

To guide personalized therapy for Tailoring immunotherapy to individual patients, reducing unnecessary toxicity and cost.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with radiologically or histologically confirmed advanced HCC
* Candidates for systemic immune checkpoint inhibitors (e.g., atezolizumab-bevacizumab, durvalumab-tremelimumab).
* Patients with preserved liver function. ( up to G2 using ALBI score or up to B (7 ) using Child-Pugh socring system) .

Exclusion Criteria:

* Child-Pugh C liver function.
* Prior liver transplantation.
* patients with concurrent malignancies other than HCC.
* Active autoimmune disease requiring systemic immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with advanced hepatocellular carcinoma either denovoor after prior line of treatment
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
ICI-Specific Survival (OS-ICI). | 12 months
  Time from ICI initiation to death or last follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Sohag university hospitals, Sohag, Sohag Governorate
  - sSohag oncology centre, Sohag, Sohag Governorate

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 10. Cheng, A. L., Rimassa, L., Ducreux, M., et al. (2022). J Hepatol, 76, 862-873.
- [Background] 9. Yau, T., Cheng, A. L., Rimassa, L., et al. (2025). Lancet, 405, 1851-1864.
- [Background] 8. Llovet, J. M., Yau, T., Cheng, A. L., et al. (2008). N Engl J Med, 359, 378-390.
- [Background] 7. Reig, M., Llovet, J. M., Yau, T., et al. (2021). J Hepatol, 76, 681-693.
- [Background] 6. Singal, A. G., Reig, M., Llovet, J. M., et al. (2023). Hepatology, 78, 1922-1965.
- [Background] El-Serag HB. Hepatocellular carcinoma: recent trends in the United States. Gastroenterology. 2004 Nov;127(5 Suppl 1):S27-34. doi: 10.1053/j.gastro.2004.09.013. PMID 15508094
- [Background] Kalligeros M, Henry L, Younossi ZM. Metabolic dysfunction-associated steatotic liver disease and its link to cancer. Metabolism. 2024 Nov;160:156004. doi: 10.1016/j.metabol.2024.156004. Epub 2024 Aug 23. PMID 39182603
- [Background] 3. Liu, Y., Kalligeros, M., El-Serag, H. B., et al. (2022). Cancer Med, 11, 1310-1323.
- [Background] 2. McGlynn, K. A., Liu, Y., Kalligeros, M., et al. (2021). Hepatology, 73, 4-13.
- [Background] 1. Siegel, R. L., McGlynn, K. A., Liu, Y., et al. (2024). CA Cancer J Clin, 74, 12-49.